CLINICAL TRIAL: NCT01829113
Title: Double-Blind Randomized Phase II Trial of Carboplatin and Pemetrexed With or Without OGX-427 in Patients With Previously Untreated Stage IV Non-Squamous-Non-Small-Cell Lung Cancer (The Spruce Clinical Trial)
Brief Title: Phase II Trial of Carboplatin and Pemetrexed +/- OGX-427 in Untreated Stage IV Non-Squamous-Non-Small-Cell Lung Cancer
Acronym: Spruce
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCRI LUN 229
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Non Squamous Non Small Cell Lung Cancer
Keywords: Recurrent Lung Cancer; Stage IV Lung Cancer; OGX-427; Sarah Cannon Research Institute; SCRI; OncoGenex; NSCLC; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — apatorsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OGX-427 (Experimental): Three loading doses of OGX-427 at 600mg intravenously (IV) will be administered over 9 days. Following the loading dose period, OGX-427 will be administered at 600mg IV weekly Days 1, 8 and 15 of each 21 day cycle during the Treatment Phase. The Treatment Phase will be followed by a Maintenance Phase of OGX-427 administered at 600mg IV weekly Days 1, 8 and 15 of each 21 day cycle.
  Interventions: Drug: OGX-427
- Placebo (Placebo Comparator): Three loading doses of placebo will be administered intravenously (IV) over 9 days. Following the loading dose period, placebo will be administered IV weekly Days 1, 8 and 15 of each 21 day cycle during the Treatment Phase. The Treatment Phase will be followed by a Maintenance Phase of placebo administered IV weekly Days 1, 8 and 15 of each 21 day cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OGX-427 — Three loading doses of 600mg OGX-427 will be administered intravenously (IV) during a 9 day period. Then 600mg IV OGX-427 will be given weekly on Days 1, 8 and 15 of each 21 day cycle prior to the administration of pemetrexed (500mg/m^2 IV) and carboplatin (AUC 6 IV) on Day 1 of each cycle for a maximum of four treatment cycles. Patients who respond to treatment or have stable disease will continue to receive 600 mg IV OGX-427 plus 500mg/m2 IV pemetrexed weekly until toxicity or disease progression.
  Other Names: apatorsen
  Arms: OGX-427
Drug: Placebo — Three loading doses of placebo will be administered intravenously (IV) during a 9 day period. Then placebo (IV) will be given weekly on Days 1, 8 and 15 of each 21 day cycle prior to the administration of pemetrexed (500mg/m^2 IV) and carboplatin (AUC 6 IV) on Day 1 of each cycle for a maximum of four treatment cycles. Patients who respond to treatment or have stable disease will continue to receive placebo (IV) plus 500mg/m2 IV pemetrexed weekly until toxicity or disease progression.
  Arms: Placebo

SUMMARY:
This randomized phase II study will compare the efficacy and safety of the combination of carboplatin and pemetrexed with and without OGX-427 in patients with previously untreated advanced non-squamous NSCLC.

DETAILED DESCRIPTION:
Modern doublet chemotherapy improves survival in patients with advanced non-small cell lung cancer (NSCLC) compared with supportive care alone, with non-squamous NSCLC patients treated with platinum/pemetrexed living longer than patients treated with platinum/gemcitabine. Despite these advances, poor outcomes with advanced disease warrant exploration of novel drugs with unique mechanisms of action. Preclinical evidence in lung cancer models shows promising antitumor activity with OGX-427 in combination with platinum based therapy or pemetrexed. In this double-blind, placebo-controlled, Phase II study, pemetrexed and carboplatin plus OGX-427 followed by maintenance pemetrexed and OGX-427 will be compared with pemetrexed and carboplatin plus placebo followed by maintenance pemetrexed and placebo in patients with previously untreated advanced non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of advanced NSCLC, excluding squamous cell and small cell histology. Tumors with mixed NSCLC histologies are eligible, as long as the predominant histology is not squamous. If small-cell elements are present or not otherwise specified histologically, the patient is not eligible.
2. Metastatic disease (according to American Joint Committee on Cancer (AJCC) staging system, v7.0).
3. No prior systemic chemotherapy, immunotherapy, targeted therapy, or biological therapy for metastatic disease; previous adjuvant or neoadjuvant therapy for Stage I, II, or III disease is allowed as long as the interval from the end of treatment until disease progression was >12 months.
4. No prior radiation therapy to the whole pelvis or to ≥25% of the total bone marrow area. Other radiation therapy must be completed at least 2 weeks prior to study entry. Must have recovered from acute adverse effects prior to study entry.
5. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
7. Baseline laboratory values as follows:

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Hemoglobin (Hgb) ≥10 g/dL
   * Platelets ≥100,000/μL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ≤3.0 x the upper limit of normal (ULN); 5 x ULN if known hepatic metastases.
   * Total bilirubin ≤1.5 x ULN, unless secondary to Gilbert's disease
   * Serum creatinine ≤1.5 x ULN. If creatinine is >1.5, calculate creatinine clearance (CrCl) ≥45 mL/min by the Cockcroft-Gault method:

   Glomerular Filtration Rate (GFR) = (140-age) x (weight/kg) x (0.85 if female)/(72 x serum creatinine mg/dL)
8. Fertile male patients willing to use adequate contraceptive measures.
9. Female patients who are not of child-bearing potential, and fertile female patients of child-bearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 72 hours prior to start of randomization.
10. Life expectancy ≥ 12 weeks.
11. Must be ≥18 years of age at the time of consent.
12. Willingness and ability to comply with trial and follow-up procedures.
13. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

1. Known anaplastic lymphoma kinase (ALK) translocation and epidermal growth factor receptor (EGFR) "activating" mutations where first-line treatment with targeted tyrosine kinase inhibitor therapy is more appropriate.
2. Known central nervous system (CNS) disease other than neurologically stable, treated brain metastases defined as metastasis having no evidence of progression or hemorrhage after treatment and no ongoing requirements for corticosteroids, (e.g., dexamethasone) for at least 2 weeks.
3. Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association (NYHA) ≥ Class 2:

   * Unstable angina pectoris
   * Congestive heart failure
   * Acute myocardial infarction
   * Conduction abnormality not controlled with pacemaker or medication
   * Significant ventricular or supraventricular arrhythmias (Patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
4. Patients currently receiving therapeutic anticoagulation.
5. Pregnant or lactating women.
6. Any serious, active underlying medical condition that would impair the ability of the patient to receive study treatment, such as diabetes mellitus or infection.
7. Unable or unwilling to take folic acid or vitamin B12.
8. Active second malignancy (except non-melanomatous skin or superficial bladder cancer) defined as requiring current need for cancer therapy or at high risk of recurrence (>30%) during the study.
9. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
10. Inability or unwillingness to comply with trial and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, M.D., Study Chair — SCRI
Locations (16):
- United States (16):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Florida Hospital Cancer Insitute, Orlando, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Baptist Hospital East, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Research Medical Center, Kansas City, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Gronberg BH, Bremnes RM, Flotten O, Amundsen T, Brunsvig PF, Hjelde HH, Kaasa S, von Plessen C, Stornes F, Tollali T, Wammer F, Aasebo U, Sundstrom S. Phase III study by the Norwegian lung cancer study group: pemetrexed plus carboplatin compared with gemcitabine plus carboplatin as first-line chemotherapy in advanced non-small-cell lung cancer. J Clin Oncol. 2009 Jul 1;27(19):3217-24. doi: 10.1200/JCO.2008.20.9114. Epub 2009 May 11. PMID 19433683
- [Background] Scagliotti GV, Parikh P, von Pawel J, Biesma B, Vansteenkiste J, Manegold C, Serwatowski P, Gatzemeier U, Digumarti R, Zukin M, Lee JS, Mellemgaard A, Park K, Patil S, Rolski J, Goksel T, de Marinis F, Simms L, Sugarman KP, Gandara D. Phase III study comparing cisplatin plus gemcitabine with cisplatin plus pemetrexed in chemotherapy-naive patients with advanced-stage non-small-cell lung cancer. J Clin Oncol. 2008 Jul 20;26(21):3543-51. doi: 10.1200/JCO.2007.15.0375. Epub 2008 May 27. PMID 18506025
- [Background] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Background] Wu R, Kausar H, Johnson P, Montoya-Durango DE, Merchant M, Rane MJ. Hsp27 regulates Akt activation and polymorphonuclear leukocyte apoptosis by scaffolding MK2 to Akt signal complex. J Biol Chem. 2007 Jul 27;282(30):21598-608. doi: 10.1074/jbc.M611316200. Epub 2007 May 17. PMID 17510053
- [Background] Zheng C, Lin Z, Zhao ZJ, Yang Y, Niu H, Shen X. MAPK-activated protein kinase-2 (MK2)-mediated formation and phosphorylation-regulated dissociation of the signal complex consisting of p38, MK2, Akt, and Hsp27. J Biol Chem. 2006 Dec 1;281(48):37215-26. doi: 10.1074/jbc.M603622200. Epub 2006 Oct 2. PMID 17015449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2013 and February 2015, a total of 155 patients (77 patients on the OGX-427 (apatorsen) arm and 78 patients on the placebo arm) were enrolled and randomized on the study.
Pre-assignment Details: Subjects were enrolled and randomized in a 1:1 ratio to receive a combination of pemetrexed and carboplatin plus either OGX-427 (apatorsen) or a placebo.
Groups:
- OGX-427: OGX-427: Three loading doses of OGX-427 at 600mg intravenously (IV) will be administered over 9 days.
  Following the loading dose period, OGX-427 will be administered at 600mg IV weekly Days 1, 8 and 15 of each 21 day cycle. OGX-427 will be given prior to the administration of pemetrexed (500mg/m2 IV) and carboplatin (AUC 6 IV) on Day 1 of each cycle. A maximum of four treatment cycles will be administered.
  Patients without toxicity or disease progression after four cycles of therapy will move on to a Maintenance Phase of OGX-427 administered at 600mg IV weekly Days 1, 8 and 15 of each 21 day cycle plus pemetrexed (500mg/m2 IV on Day 1). Patients may remain on maintenance as long as they are benefiting and have no evidence of disease progression.
- Placebo: Placebo: Three loading doses of placebo will be administered intravenously (IV) over 9 days.
  Following the loading dose period, placebo will be administered IV weekly Days 1, 8 and 15 of each 21 day cycle. Placebo will be given prior to the administration of pemetrexed (500mg/m2 IV) and carboplatin (AUC 6 IV) on Day 1 of each cycle. A maximum of four treatment cycles will be administered.
  Patients without toxicity or disease progression after four cycles of therapy will move on to a Maintenance Phase of placebo administered IV weekly Days 1, 8 and 15 of each 21 day cycle plus pemetrexed (500mg/m2 IV on Day 1). Patients may remain on maintenance as long as they are benefiting and have no evidence of disease progression.
Period: Overall Study
Arm/Group | OGX-427 | Placebo
Started | 77 (Three patients were enrolled and randomized but never received treatment.) | 78 (Two patients were enrolled and randomized but never received treatment.)
Completed | 0 | 0
Not Completed | 77 | 78
Not completed — Disease Progression | 37 | 48
Not completed — Adverse Event | 14 | 10
Not completed — Withdrawal by Subject | 17 | 10
Not completed — Death | 4 | 6
Not completed — Sponsor Decision | 1 | 1
Not completed — No Study Treatment Received | 3 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Patients that were randomized to either OGX-427 or placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | OGX-427 | Placebo | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 29 | 64
  >=65 years | 42 | 49 | 91
Age, Continuous [Median (Full Range); unit: years] | 66 [32 to 82] | 67 [38 to 82] | 66 [32 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 38 | 38 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 3 | 13
  White | 67 | 74 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77 | 78 | 155

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival
Description: Defined as the time (in months) from date of randomization to the date of first observation of progression based on radiological assessment by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1, or date of death from any cause, in the absence of progressive disease (PD) or censored at the date of last adequate tumor assessment. Progressive Disease is defined by RECIST v1.1 as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest (nadir) sum while on study (this includes the baseline sum if that is the smallest on study), or the appearance of one or more new lesions.
Time Frame: Every 6 weeks for up to 24 months
Population: All patients who were randomized
Measure: Median (95% Confidence Interval); unit: months
Groups:
- OGX-427: OGX-427: Three loading doses of OGX-427 at 600mg IV will be administered Days -9 to -1.
  Following the loading dose period, OGX-427 will be administered at 600mg IV weekly Days 1, 8 and 15 of each 21 day cycle during the Treatment Phase. OGX-427 will be given prior to the administration of pemetrexed (500mg/m2 IV) and carboplatin (AUC 6 IV) on Day 1 of each cycle. A maximum of four treatment cycles will be administered.
  Patients with objective response or stable disease after four cycles of therapy will move on to a Maintenance Phase of OGX-427 administered at 600mg IV weekly Days 1, 8 and 15 of each 21 day cycle plus pemetrexed (500mg/m2 IV on Day 1). Patients may remain on maintenance as long as they are benefiting and have no evidence of disease progression.
- Placebo: Placebo: Three loading doses of placebo will be administered IV Days -9 to -1.
  Following the loading dose period, placebo will be administered IV weekly Days 1, 8 and 15 of each 21 day cycle during the Treatment Phase. Placebo will be given prior to the administration of pemetrexed (500mg/m2 IV) and carboplatin (AUC 6 IV) on Day 1 of each cycle. A maximum of four treatment cycles will be administered.
  Patients with objective response or stable disease after four cycles of therapy will move on to a Maintenance Phase of placebo administered IV weekly Days 1, 8 and 15 of each 21 day cycle plus pemetrexed (500mg/m2 IV on Day 1). Patients may remain on maintenance as long as they are benefiting and have no evidence of disease progression.
Arm/Group | OGX-427 | Placebo
Number analyzed (Participants) | 77 | 78
months | 6 [3.3 to 8] | 4.9 [4.4 to 5.9]

2. Secondary Outcome: Number of OGX-427 Versus Placebo Participants With an Objective Response
Description: Defined as the number of patients with objective evidence of complete or partial response (CR or PR) using RECIST v 1.1. A CR is the complete disappearance of all target lesions. A PR is a decrease in baseline of 30% or more of the diameter(s) of all target lesions.
Time Frame: Every 6 weeks for up to 24 months
Population: All patients who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | OGX-427 | Placebo
Number analyzed (Participants) | 77 | 78
Participants | 21 | 25

3. Secondary Outcome: Median Overall Survival
Description: Defined as the time (in months) from date of randomization to date of death from any cause, or censored at the date last known alive.
Time Frame: Every 6 weeks for up to 41 months
Population: All patients who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | OGX-427 | Placebo
Number analyzed (Participants) | 77 | 78
Months | 10.8 [8.9 to 14.8] | 11.8 [8.0 to 16.1]

4. Secondary Outcome: Number of Patients With a Treatment-Related Adverse Event as a Measure of Safety.
Description: A treatment-related adverse event was any untoward medical occurrence in a participant which was considered to have a relationship with the study drug (suspected to be possibly or probably related to the study drug per the Investigator's assessment). Adverse events were evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Time Frame: Weekly during each 21 days cycle and for 30 days after last dose for up to 29 Months
Population: Randomized patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | OGX-427 | Placebo
Number analyzed (Participants) | 74 | 76
Participants | 63 | 70

ADVERSE EVENTS:
Time Frame: Weekly during each 21 days cycle and for 30 days after last dose for up to 29 Months
Description: Any untoward medical occurrence in a participant regardless of the relationship with the study drug per the Investigator's assessment. Adverse events were evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. All-Cause Mortality was assessed in all randomized participants, while Serious and Other (Not Including Serious) Adverse Events was only assessed in participants who received at least one dose of study treatment.
Arm/Group | OGX-427 | Placebo
All-Cause Mortality (participants affected / at risk) | 56/77 | 61/78
Serious Adverse Events (participants affected / at risk) | 35/74 | 32/76
Other Adverse Events (participants affected / at risk) | 72/74 | 75/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OGX-427 (N=74) | Placebo (N=76)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Arteriosclerosis (Vascular disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Death (General disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OGX-427 (N=74) | Placebo (N=76)
Fatigue (General disorders) | 46 | 50
Nausea (Gastrointestinal disorders) | 44 | 44
Anaemia (Blood and lymphatic system disorders) | 41 | 47
Constipation (Gastrointestinal disorders) | 37 | 34
Skin and subcutaneous tissue disorders (Metabolism and nutrition disorders) | 35 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 32 | 30
Vomiting (Gastrointestinal disorders) | 28 | 24
Diarrhoea (Gastrointestinal disorders) | 27 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 21
Neutropenia (Blood and lymphatic system disorders) | 23 | 36
Decreased appetite (Metabolism and nutrition disorders) | 21 | 20
Oedema peripheral (General disorders) | 17 | 15
Dizziness (Nervous system disorders) | 16 | 16
Dehydration (Metabolism and nutrition disorders) | 14 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 31
Pyrexia (General disorders) | 13 | 11
Asthenia (General disorders) | 12 | 11
Insomnia (Psychiatric disorders) | 12 | 18
Leukopenia (Blood and lymphatic system disorders) | 12 | 20
Weight decreased (Investigations) | 12 | 10
Chills (General disorders) | 11 | 4
Abdominal pain (Gastrointestinal disorders) | 10 | 8
Chest pain (General disorders) | 10 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 12
Anxiety (Psychiatric disorders) | 9 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 13
Hypotension (Vascular disorders) | 9 | 10
Paraesthesia (Nervous system disorders) | 9 | 6
Platelet count decreased (Investigations) | 9 | 10
Urinary tract infection (Infections and infestations) | 9 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 0
Mucosal inflammation (General disorders) | 8 | 11
Pneumonia (Infections and infestations) | 8 | 7
Rash (Metabolism and nutrition disorders) | 8 | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Fall (Injury, poisoning and procedural complications) | 7 | 4
Lacrimation increased (Eye disorders) | 7 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 11
Alanine aminotransferase increased (Investigations) | 6 | 7
Aspartate aminotransferase increased (Investigations) | 6 | 7
Blood creatinine increased (Investigations) | 6 | 4
Dysgeusia (Nervous system disorders) | 6 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Night sweats (Metabolism and nutrition disorders) | 6 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Headache (Nervous system disorders) | 5 | 15
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Pain (General disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 8
Stomatitis (Gastrointestinal disorders) | 5 | 6
White blood cell count decreased (Investigations) | 5 | 8
Blood alkaline phosphatase increased (Investigations) | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 4
Dry skin (Metabolism and nutrition disorders) | 4 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 2
Flushing (Vascular disorders) | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4
Hot flush (Vascular disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 7
Hypertension (Vascular disorders) | 4 | 15
Neuropathy peripheral (Nervous system disorders) | 4 | 7
Neutrophil count decreased (Investigations) | 4 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Sinusitis (Infections and infestations) | 4 | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Depression (Psychiatric disorders) | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 11
Hyperhidrosis (Metabolism and nutrition disorders) | 3 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5
Rash maculo-papular (Metabolism and nutrition disorders) | 3 | 7
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Vision blurred (Eye disorders) | 3 | 5
Candida infection (Infections and infestations) | 2 | 4
Confusional state (Psychiatric disorders) | 2 | 4
Dry eye (Eye disorders) | 2 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Malaise (General disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Tachycardia (Cardiac disorders) | 2 | 6
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Bronchitis (Infections and infestations) | 1 | 4
Deep vein thrombosis (Vascular disorders) | 1 | 6
Conjunctivitis (Infections and infestations) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2014-11-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT01829113/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT01829113/SAP_001.pdf